CLINICAL TRIAL: NCT02054247
Title: The Placebo-Controlled Continuous And Pulsed Ultrasound Treatments on Carpal Tunnel Syndrome : A Randomised Trial
Brief Title: Continuous And Pulsed Ultrasound Treatments On Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Onur Armağan, Onur Armagan MD, Eskisehir Osmangazi University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: clinics-2013-0627
Record Dates: First submitted 2014-01-27; First posted 2014-02-04 (Estimated); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal tunnel syndrome,ultrasound,pulsed ultrasound
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ultrasound (Experimental): ultrasound : a frequency of 1 megahertz and with an intensity of 1 W/cm2
  Interventions: Device: ultrasound
- pulsed ultrasound (Experimental): pulsed ultrasound : a frequency of 1 megahertz and with an intensity of 1 W/cm2 and a pulsed mode duty cycle of 1:4
  Interventions: Device: pulsed ultrasound
- placebo ultrasound (Placebo Comparator): placebo ultrasound : same ultrasound device as described above seemed to be working but without delivering any output
  Interventions: Device: placebo ultrasound

INTERVENTIONS:
Device: ultrasound — a frequency of 1 megahertz and with an intensity of 1 W/cm2, 5 days a week for a total of 15 sessions
  Arms: ultrasound
Device: pulsed ultrasound — a frequency of 1 megahertz and with an intensity of 1 W/cm2 and a pulsed mode duty cycle of 1:4, 5 days a week for a total of 15 sessions
  Arms: pulsed ultrasound
Device: placebo ultrasound — same ultrasound device as described above seemed to be working but without delivering any output, 5 days a week for a total of 15 sessions
  Arms: placebo ultrasound

SUMMARY:
The aim of this placebo-controlled study was to evaluate the effects of pulsed and continuous ultrasound treatments combined with splint therapy on patients with mild and moderate idiopathic carpal tunnel syndrome

DETAILED DESCRIPTION:
The study included 36 carpal tunnel syndrome patients who were randomly divided into 3 groups.The first group received 0 W/cm2 placebo ultrasound treatment. second group received 1.0 W/cm2 continuous ultrasound treatment and the third group received 1.0 W/cm2 1:4 pulsed ultrasound treatment 5 days a week for a total of 15 sessions. All patients were also treated with night splints during the treatment. Pretreatment and posttreatment Visual Analogue Scale scores, Symptom Severity Scale scores, Functional Status Scale scores, median nerve motor conduction velocity. and distal latency and sensory conduction velocity of median nerve in the 2nd finger and palm were compared.

ELIGIBILITY:
Inclusion Criteria:

* Mild or moderate idiopathic carpal tunnel syndrome (without thenar atrophy or spontaneous activity on electrophysiological examination of the abductor pollicis brevis (APB) muscle)

Exclusion Criteria:

* Secondary entrapment neuropathies
* Cervical radiculopathy
* Systemic diseases with increased risk of the carpal tunnel syndrome
* Gained surgical relief of the syndrome
* Treated with ultrasound for the syndrome
* A history of steroid injections into the carpal tunnel and of physical therapy within the last 3 months
* Patients with either thenar atrophy or spontaneous activity (fibrillation potentials and positive sharp waves) on electrophysiological examination

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Onur ARMAGAN, ass. prof., Study Director — Eskisehir Osmangazi University

REFERENCES:
- [Derived] Armagan O, Bakilan F, Ozgen M, Mehmetoglu O, Oner S. Effects of placebo-controlled continuous and pulsed ultrasound treatments on carpal tunnel syndrome: a randomized trial. Clinics (Sao Paulo). 2014 Aug;69(8):524-8. doi: 10.6061/clinics/2014(08)04. PMID 25141110

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrasound | Pulsed Ultrasound | Placebo Ultrasound
Started | 15 | 16 | 15
Completed | 15 | 16 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasound | Pulsed Ultrasound | Placebo Ultrasound | Total
Number analyzed (Participants) | 15 | 16 | 15 | 46
Age, Continuous [Mean (Standard Deviation); unit: years]
  age mean | 43.31 (2.79) | 45.20 (2.98) | 44.53 (2.38) | 44.34 (2.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 15 | 46
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 15 | 16 | 15 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Symptom Severity With Symptom Severity Scale
Description: Post treatment comparison of Symptom Severity Scale between three groups minimum score is 11, maximum score is 55. The clinic of patient worses when the score increases.
Time Frame: three weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ultrasound | Pulsed Ultrasound | Placebo Ultrasound
Number analyzed (Participants) | 15 | 16 | 15
units on a scale | 23.06 (8.13) | 22.06 (8.73) | 19.66 (4.60)
Statistical Analysis 1: Comparison: Ultrasound vs Pulsed Ultrasound vs Placebo Ultrasound; Test type: Superiority; p = 0.442, ANOVA

2. Secondary Outcome: Change From Baseline in Pain With Visual Analogue Scale
Description: Post treatment comparison of Visual Analogue Scale between three groups min score is 0, maximum score is 10. The clinic of patient worses when the score increases.
Time Frame: Three weeks
Population: ultrasound group has 15, pulsed us group has 16, placebo us group has 15 patients
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Ultrasound | Pulsed Ultrasound | Placebo Ultrasound
Number analyzed (Participants) | 15 | 16 | 15
score | 4.40 (2.32) | 2.68 (1.92) | 3.53 (1.95)
Statistical Analysis 1: Comparison: Ultrasound vs Pulsed Ultrasound vs Placebo Ultrasound; Test type: Superiority; p = 0.083, ANOVA

3. Secondary Outcome: Change From Baseline in Functional Status With Functional Status Scale
Description: Post treatment comparison of Functional Status Scale between three groups min score is 8, maximum score is 40. The clinic of patient worses when the score increases.
Time Frame: Three weeks
Population: ultrasound group has 15 patients, pulsed us group has 16 patients, placebo us has 15 patients.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Ultrasound | Pulsed Ultrasound | Placebo Ultrasound
Number analyzed (Participants) | 15 | 16 | 15
score | 18.8 (7.34) | 19.31 (9.42) | 14.2 (4.52)
Statistical Analysis 1: Comparison: Ultrasound vs Pulsed Ultrasound vs Placebo Ultrasound; Test type: Superiority; p = 0.125, ANOVA

4. Secondary Outcome: Changes From Baseline Nervus Medianus Motor Conduction Velocity
Description: Post treatment comparison of Median motor nerve conduction velocity between three groups
Time Frame: Three weeks
Population: ultrasound group has 15 patients, pulsed us group has 16 patients, placebo us group has 15 patients.
Measure: Mean (Standard Deviation); unit: meter/seconds
Arm/Group | Ultrasound | Pulsed Ultrasound | Placebo Ultrasound
Number analyzed (Participants) | 15 | 16 | 15
meter/seconds | 54.26 (4.29) | 55.68 (5.24) | 57.91 (5.44)
Statistical Analysis 1: Comparison: Ultrasound vs Pulsed Ultrasound vs Placebo Ultrasound; Test type: Superiority; p = 0.146, ANOVA

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Ultrasound | Pulsed Ultrasound | Placebo Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No